CLINICAL TRIAL: NCT04452435
Title: A Randomised, Double-blind, Placebo-controlled, Phase 2 Trial Investigating the Safety and Efficacy of C21 in Hospitalised Subjects With COVID-19 Infection Not Requiring Mechanical Ventilation
Brief Title: Safety and Efficacy of C21 in Subjects With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vicore Pharma AB (Industry)
Collaborators: Orphan Reach Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VP-C21-006; 2020-001502-38 (EudraCT Number)
Record Dates: First submitted 2020-06-29; First posted 2020-06-30 (Actual); Results first posted 2021-04-30 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: COVID-19
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — compound 21

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C21 100 mg twice daily (Experimental): Oral C21 treatment 100 mg twice daily for 7 days
  Interventions: Drug: C21
- Placebo (Placebo Comparator): Oral placebo treatment 100 mg twice daily for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: C21 — C21
  Arms: C21 100 mg twice daily
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a randomised, double-blind, placebo-controlled phase 2 trial investigating the safety and efficacy of C21 in subjects who are hospitalised with COVID-19 infection, but not in need of mechanical invasive or non-invasive ventilation.

In total, approximately 100 subjects will be enrolled and randomised to receive twice daily oral administration of either standard of care (SoC) + placebo (N=50) or SoC + C21 (N=50). Subjects will be treated for 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent, consistent with ICH-GCP R2 and local laws, obtained before the initiation of any trial related procedure
2. Diagnosis of coronavirus (SARS-CoV)-2 infection confirmed by polymerase chain reaction (PCR) test < 4 days before Visit 1 with signs of an acute respiratory infection
3. Age > 18 and < 70 years
4. CRP > 50 and < 150 mg/l
5. Admitted to a hospital or controlled facility (home quarantine is not sufficient)
6. In the opinion of the Investigator, the subject will be able to comply with the requirements of the protocol

Exclusion Criteria:

1. Any previous experimental treatment for COVID-19
2. Need for mechanical invasive or non-invasive ventilation
3. Concurrent respiratory disease such as COPD (chronic obstructive pulmonary disease), IPF and/or intermittent, persistent or more severe asthma requiring daily therapy or any subjects that have had an asthma flare requiring corticosteroids in the 4 weeks (28 days) prior to COVID-19 diagnosis
4. Participation in any other interventional trial within 3 months prior to Visit 1
5. Any of the following findings at Visit 1:

   * Positive results for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCVAb) or human immunodeficiency virus 1+2 antigen/antibody (HIV 1+2 Ag/Ab
   * Positive pregnancy test (see Section 8.2.3)
6. Clinically significant abnormal laboratory value at Visit 1 indicating a potential risk for the subject if enrolled in the trial as evaluated by the Investigator
7. Concurrent serious medical condition with special attention to cardiac or ophthalmic conditions (e.g. contraindications to cataract surgery), which in the opinion of the Investigator makes the subject inappropriate for this trial
8. Malignancy within the past 3 years with the exception of in situ removal of basal cell carcinoma and cervical intraepithelial neoplasia grade I
9. Treatment with any of the medications listed below within 1 week prior to Visit 1:

   1. Strong Cytochrome p450 (CYP) 3A4 inducers (e.g. rifampicin, phenytoin, St. John's Wort, phenobarbital, rifabutin, carbamazepine, anti HIV drugs, barbiturates)
   2. Warfarin
10. Pregnant or breast-feeding female subjects
11. Female subjects of childbearing potential not willing to use contraceptive methods as described in Section 5.3.1
12. Male subjects not willing to use contraceptive methods as described in Section 5.3.1
13. Subjects known or suspected of not being able to comply with this trial protocol (e.g. due to alcoholism, drug dependency or psychological disorder)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2020-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Porter, MD, Principal Investigator — Respiratory Medicine, University College Hospital
Locations (9):
- India (8):
  - Department of Medicine, Civil Hospital and B J Medical College, Ahmedabad, Gujarat
  - Infectious Disease, Metas Adventist Hospital, Surat, Gujarat
  - Clinical Research Department, Basement, Unity Trauma Centre and ICU (Unity Hospital, Surat, Gujarat
  - First Floor Clinical Research Department Rhythm Heart Institute, Vadodara, Gujarat
  - Internal Medicine S.L. Raheja Hospital, Mumbai, Maharashtra
  - Department of Medicine, Government Medical College and Hospital, Nagpur, Maharashtra
  - Neuro Critical Care, Grant Medical Foundation Ruby Hall Clinic, Pune, Maharashtra
  - Department of Medicine, Noble Hospitals Pvt. Ltd, Pune, Maharashtra
- Respiratory Medicine, University College Hospital, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 96 enrolled subjects were screening failures because inclusion criteria 4 was not met.
  2 enrolled subjects decided to withdraw from the trial before randomization. 2 subjects died before randomization (pneumonia). The remaining 106 subjects were randomized to trial treatment.
Groups:
- C21 Treatment: Oral C21 treatment 100 mg twice daily for 7 days
- Placebo Treatment: Oral placebo treatment twice daily for 7 days
Period: Screening
Arm/Group | C21 Treatment | Placebo Treatment
Started | 51 | 55
Completed | 51 | 55
Not Completed | 0 | 0
Period: Treatment Period
Arm/Group | C21 Treatment | Placebo Treatment
Started | 51 | 55
Completed | 45 | 43
Not Completed | 6 | 12
Period: Follow-up
Arm/Group | C21 Treatment | Placebo Treatment
Started | 45 | 43
Completed | 45 | 42
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | C21 Treatment | Placebo Treatment | Total
Number analyzed (Participants) | 51 | 55 | 106
Age, Continuous [Mean (Full Range); unit: years] | 54.3 [29 to 68] | 51.1 [22 to 68] | 52.6 [22 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 38 | 42 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 51 | 55 | 106
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 51 | 55 | 106
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  India | 51 | 55 | 106
Height [Mean (Full Range); unit: cm] | 166.1 [132 to 198] | 166.0 [143 to 188] | 166.1 [132 to 198]
Weight [Mean (Full Range); unit: kg] | 70.1 [46 to 116] | 69.2 [47 to 112] | 69.6 [46 to 116]
Body mass index [Mean (Full Range); unit: kg/m^2] | 25.4 [15 to 41] | 25.1 [20 to 34] | 25.2 [15 to 41]
Supplemental oxygen use at baseline [Count of Participants; unit: Participants] — Number of subjects in use of supplemental oxygen use at baseline
  Participants | 29 | 32 | 61
CRP value ≤ median [Count of Participants; unit: Participants] — Number of subjects with baseline CRP value ≤ median
  Participants | 24 | 22 | 46
CRP value > median [Count of Participants; unit: Participants] — Number of subjects with baseline CRP value > median
  Participants | 21 | 25 | 46

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in C-reactive Protein (CRP) After Treatment With C21 200 mg Daily Dose (100 mg b.i.d.)
Description: Change in C-reactive protein (CRP) from baseline to the average of the last two assessments in the treatment period
Time Frame: Treatment period of 7 days (Day 1 to Day 8)
Population: Full analysis set. A total of 45 subjects in the C21 group and 46 subjects in the placebo group were included in the analysis of the primary endpoint in the FAS. For a number of the excluded subjects, the reason for exclusion from the primary endpoint analysis was that they had no baseline value available.
Measure: Least Squares Mean (90% Confidence Interval); unit: mg/L
Arm/Group | C21 Treatment | Placebo Treatment
Number analyzed (Participants) | 45 | 46
mg/L | 0.19 [0.14 to 0.25] | 0.22 [0.17 to 0.29]
Statistical Analysis 1: Comparison: C21 Treatment vs Placebo Treatment; Test type: Equivalence — The null hypothesis was that the treatments were equivalent and was to be rejected in favour of the alternative hypothesis that a treatment difference existed, if the probability of the null hypothesis being true was less than 10%; p = 0.4891, ANCOVA
Statistical Analysis 2: Comparison: C21 Treatment vs Placebo Treatment; A subgroup analyses was performed in subjects with supplemental oxygen use at baseline. A total of 26 subjects in the C21 group and 27 in the placebo group were included in the analysis of change in CRP from baseline to the mean of the last 2 non-missing scheduled assessments during the treatment period by baseline supplemental oxygen use; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0881, ANCOVA

2. Secondary Outcome: Change From Baseline in Body Temperature
Description: Change in body temperature from baseline to the average of the last two assessments in the treatment period
Time Frame: Treatment period of 7 days ((Day 1 to Day 8)
Population: Subjects with measurements were included in the analysis for the full analysis set.
Measure: Least Squares Mean (90% Confidence Interval); unit: °C
Arm/Group | C21 Treatment | Placebo Treatment
Number analyzed (Participants) | 51 | 54
°C | -0.11 [-0.25 to 0.02] | -0.34 [-0.47 to -0.21]
Statistical Analysis 1: Comparison: C21 Treatment vs Placebo Treatment; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0492, ANCOVA

3. Secondary Outcome: Change From Baseline in IL-6
Description: Change in IL-6 from baseline to the average of the last two assessments during the treatment period
Time Frame: Treatment period of 7 days (Day 1 to Day 8)
Population: Subjects with measurements were included in the analysis for the full analysis set.
Measure: Least Squares Mean (90% Confidence Interval); unit: pg/mL
Arm/Group | C21 Treatment | Placebo Treatment
Number analyzed (Participants) | 31 | 34
pg/mL | 0.73 [0.51 to 1.05] | 0.73 [0.51 to 1.03]
Statistical Analysis 1: Comparison: C21 Treatment vs Placebo Treatment; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.9923, ANCOVA

4. Secondary Outcome: Change From Baseline in IL-10
Description: Change in IL-10 from baseline to the average of the last two assessments during the treatment period
Time Frame: Treatment period of 7 days (Day 1 to Day 8)
Population: Subjects with measurements were included in the analysis for the full analysis set.
Measure: Least Squares Mean (90% Confidence Interval); unit: pg/mL
Arm/Group | C21 Treatment | Placebo Treatment
Number analyzed (Participants) | 37 | 39
pg/mL | 0.66 [0.54 to 0.8] | 0.73 [0.6 to 0.89]
Statistical Analysis 1: Comparison: C21 Treatment vs Placebo Treatment; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.5355, ANCOVA

5. Secondary Outcome: Change From Baseline in TNF
Description: Change in TNF from baseline to the average of the last two assessments during the treatment period.
Time Frame: Treatment period of 7 days (Day 1 to Day 8)
Population: Subjects with measurements were included in the analysis for the full analysis set.
Measure: Least Squares Mean (90% Confidence Interval); unit: pg/mL
Arm/Group | C21 Treatment | Placebo Treatment
Number analyzed (Participants) | 46 | 46
pg/mL | 0.91 [0.77 to 1.07] | 1.01 [0.86 to 1.19]
Statistical Analysis 1: Comparison: C21 Treatment vs Placebo Treatment; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.4738, ANCOVA

6. Secondary Outcome: Change From Baseline in CA125
Description: Change in CA125 from baseline to the average of the last two assessments in the treatment period
Time Frame: Treatment period of 7 days (Day 1 to Day 8)
Population: Subjects with measurements were included in the analysis for the full analysis set.
Measure: Least Squares Mean (90% Confidence Interval); unit: u/mL
Arm/Group | C21 Treatment | Placebo Treatment
Number analyzed (Participants) | 46 | 48
u/mL | 1.16 [1.04 to 1.31] | 1.17 [1.05 to 1.31]
Statistical Analysis 1: Comparison: C21 Treatment vs Placebo Treatment; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.9418, ANCOVA

7. Secondary Outcome: Change From Baseline in Ferritin
Description: Change in Ferritin from baseline to the average of the last two assessments during the treatment period.
Time Frame: Treatment period of 7 days (Day 1 to Day 8)
Population: Subjects with measurements were included in the analysis for the full analysis set.
Measure: Least Squares Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | C21 Treatment | Placebo Treatment
Number analyzed (Participants) | 46 | 47
ng/mL | 0.75 [0.66 to 0.84] | 0.74 [0.66 to 0.84]
Statistical Analysis 1: Comparison: C21 Treatment vs Placebo Treatment; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.9733, ANCOVA

8. Secondary Outcome: Number of Subjects Not in Need of Oxygen Supply
Description: Number of subjects not in need of oxygen supply at the end of treatment
Time Frame: End-of treatment, Day 7 or 8
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | C21 Treatment | Placebo Treatment
Number analyzed (Participants) | 51 | 55
Participants | 37 | 30
Statistical Analysis 1: Comparison: C21 Treatment vs Placebo Treatment; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0568, Regression, Logistic

9. Secondary Outcome: Number of Subjects Not in Need of Mechanical Invasive or Non-invasive Ventilation
Description: Number of subjects not in need of mechanical invasive or non-invasive ventilation during the treatment period
Time Frame: Treatment period of 7 days (Day 1 to Day 8)
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | C21 Treatment | Placebo Treatment
Number analyzed (Participants) | 51 | 55
Participants | 50 | 53
Statistical Analysis 1: Comparison: C21 Treatment vs Placebo Treatment; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.6088, Regression, Logistic

10. Secondary Outcome: Time to Need of Mechanical Invasive or Non-invasive Ventilation
Description: Time to need of mechanical invasive or non-invasive ventilation during treatment period
Time Frame: Treatment period of 7 days
Population: Subjects with measurements were included in the analysis for the full analysis set.
Measure: Mean (Full Range); unit: hours
Arm/Group | C21 Treatment | Placebo Treatment
Number analyzed (Participants) | 1 | 2
hours | 60.0 [60.0 to 60.0] | 77.925 [59.98 to 95.87]
Statistical Analysis 1: Comparison: C21 Treatment vs Placebo Treatment; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.5757, Log Rank

11. Secondary Outcome: Time on Oxygen Supply (for Those Not Needing Mechanical Invasive or Non-invasive Ventilation)
Description: Time on oxygen supply during the treatment period (for those not needing mechanical invasive or non-invasive ventilation)
Time Frame: Treatment period of 7 days (Day 1 to Day 8)
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | C21 Treatment | Placebo Treatment
Number analyzed (Participants) | 51 | 55
days | 5.0 [1.0 to 7.0] | 5.0 [1.0 to 7.0]
Statistical Analysis 1: Comparison: C21 Treatment vs Placebo Treatment; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.8588, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Adverse Events
Description: Adverse events were reported from signing of informed consent until end-of-trial visit. No AEs were reported from signing of informed consent until randomization, except for 2 fatal SAEs described under Adverse events.
Time Frame: Day 1 to end-of-trial (Visit 9)
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | C21 Treatment | Placebo Treatment
Number analyzed (Participants) | 51 | 55
Participants | 31 | 37

13. Post Hoc Outcome: Oxygen Supplementation at Day 14
Description: Number of subjects requiring oxygen supplementation at Day 14
Time Frame: Follow-up Day 14 (7 days after end-of-treatment)
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | C21 Treatment | Placebo Treatment
Number analyzed (Participants) | 51 | 55
Participants | 1 | 11
Statistical Analysis 1: Comparison: C21 Treatment vs Placebo Treatment; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.003, Chi-squared

ADVERSE EVENTS:
Time Frame: From signing of informed consent until end-of-trial visit, 14-19 days.
Description: At each visit, the subject was asked about AEs in an objective manner, e.g., "Have you experienced any problems since the last visit?" No AEs were reported from signing of informed consent until randomization except for 2 fatal SAEs.
Groups:
- No Treatment (Before Randomization): Subjects that were enrolled in the trial but not randomized
Arm/Group | C21 Treatment | Placebo Treatment | No Treatment (Before Randomization)
All-Cause Mortality (participants affected / at risk) | 1/51 | 3/55 | 2/100
Serious Adverse Events (participants affected / at risk) | 1/51 | 3/55 | 2/100
Other Adverse Events (participants affected / at risk) | 30/51 | 36/55 | 0/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | C21 Treatment (N=51) | Placebo Treatment (N=55) | No Treatment (Before Randomization) (N=100)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) — The events had a fatal outcome
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) — The events had a fatal outcome
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | C21 Treatment (N=51) | Placebo Treatment (N=55) | No Treatment (Before Randomization) (N=100)
Aspartate aminotransferase increased (Investigations) | 6 (6) | 3 (4) | NA
Blood glucose increased (Investigations) | 5 (7) | 3 (3) | NA
Interleukin level increased (Investigations) | 4 (6) | 4 (4) | NA
Alanine aminotransferase increased (Investigations) | 3 (3) | 4 (5) | NA
Serum ferritin increased (Investigations) | 5 (5) | 2 (2) | NA
Alpha tumour necrosis factor increased (Investigations) | 1 (1) | 3 (3) | NA
Carbohydrate antigen 125 increased (Investigations) | 0 (0) | 4 (4) | NA
Lymphocyte count decreased (Investigations) | 1 (1) | 3 (4) | NA
Neutrophil count increased (Investigations) | 1 (1) | 3 (5) | NA
Platelet count decreased (Investigations) | 1 (1) | 3 (3) | NA
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 2 (2) | NA
Blood calcium decreased (Investigations) | 1 (1) | 2 (2) | NA
Blood potassium increased (Investigations) | 1 (1) | 2 (2) | NA
White blood cell count increased (Investigations) | 0 (0) | 3 (4) | NA
Blood urea increased (Investigations) | 0 (0) | 2 (2) | NA
Platelet count increased (Investigations) | 0 (0) | 2 (2) | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 11 (14) | 4 (5) | NA
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | NA
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | NA
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (4) | NA
Glycosuria (Renal and urinary disorders) | 1 (1) | 3 (3) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/35/NCT04452435/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT04452435/SAP_001.pdf